CLINICAL TRIAL: NCT02967575
Title: Triadyme-C, a Polycrystalline Diamond Compact Cervical Disc Replacement (cTDR): Evaluation of Clinical and Radiographic Outcome
Brief Title: Triadyme-C, a Polycrystalline Diamond Compact Cervical Disc Replacement (cTDR)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dymicron (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP 16/01
Record Dates: First submitted 2016-11-15; First posted 2016-11-18 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Intervertebral Disc Disorder Cervical
Keywords: cervical total disc replacement (cTDR)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1- or 2-level cTDR: patients suffering from intractable symptomatic cervical disc disease (SCDD) requiring 1- or 2-level reconstruction of the disc from C3-C7
  Interventions: Device: cTDR

INTERVENTIONS:
Device: cTDR — The surgical procedure for the Triadyme-C total disc replacement corresponds to the standard surgical technique for cTDR:
  * Implantation through a standard anterior cervical approach
  * Midline identification
  * Routine discectomy with endplate preparation and decompression
  * Implant sizing and trial implantation
  * Keel preparation
  * Implant preparation and loading of the appropriate Triadyme-C implant
  * Triadyme-C insertion, positioned as close to the midline as possible
  Other Names: cervical Total Disc Replacement

SUMMARY:
This Post Market Clinical Follow-up (PMCF) is conducted to collect clinical and radiographic outcome information on patients suffering from intractable symptomatic cervical disc disease requiring 1- or 2-level reconstruction of the disc from C3-C7, after being treated with the Triadyme-C polycrystalline diamond compact cervical disc replacement.

DETAILED DESCRIPTION:
Approximately fifty percent of the population has evidence of degenerative changes in their cervical spine by the age of fifty. As part of the aging process, the intervertebral discs wear out. They lose their flexibility and elasticity and begin to collapse or even herniate. This process may result in a pathological condition called cervical Degenerative Disc Diseases (cDDD). cDDD can either be asymptomatic or symptomatic, showing different symptoms such as neck, shoulder, head, arm or leg pain, possibly associated with numbness, tingling or weakness in the upper extremity. In most cases symptomatic cDDD is initially treated conservatively with rest, immobilization, physical therapy, chiropractic manipulation and pain medication. For those cases not responding to conservative therapy, anterior cervical discectomy and fusion (ACDF) is a standard technique. The primary purpose of ACDF is to excise any disc material (discectomy), which compresses the spinal nerve or cord causing pain, sensory disturbance or weakness at the affected level, followed by interbody fusion of the adjacent vertebrae using grafts or intersomatic devices to compensate the instability and the loss of disc height resulting from discectomy. Despite the success of this common procedure, some disadvantages are to be mentioned including donor site morbidity when autografts are used, graft or device subsidence or pseudarthrosis of the segment to be fused. Besides this, physiological motion of successfully fused segments is no longer possible. This alters the loading and kinematics of adjacent spine segments which is believed by some authors to lead to adjacent segment overload as reported by several clinical and biomechanical studies. To address the disadvantages of ACDF, cervical total disc replacement (cTDR) has been developed in the 1990s, with the aim to carry the load and restore the normal disc height while preserving almost physiological segmental motion.

Today, several different cTRD designs are on the market, some of them with mid- to long-term results. A number of randomized controlled trials indicate clinical equivalence or even superiority of cTDR in some aspects compared to ACDF.

The Dymicron Triadyme-C cTDR is a two-piece articulating artificial disc prosthesis. Its patented tri-lobe articulation mechanism consists of three spherical lobes mating to three non-congruent, spherical pockets. The motion of these three lobes within their associated pockets emulates and controls natural motion of the cervical spine motion segment in all degrees of freedom.Triadyme-C is a self-centering device. This is achieved by the implant growing in height as it moves away from its center. The further away from center, the tighter the ligaments will be stretched. Each half of the Triadyme-C is a sintered monobloc, consisting of a polycrystalline diamond (PCD) bearing surface with a base of titanium-titanium carbide (Ti-TiC) composite. PCD is a sintered material composed of fused diamond crystals (typically more than 90%) and a small amount of catalyst sintering metal. The polycrystalline structure of diamond, together with the small amount of residual metal alloy, contributes significantly to the extraordinary toughness and abrasion-resistance of the material. PCD retains many of the phenomenal properties of natural diamond, including hardness, but in an isotropic form that is far more resistant to fracture.

This Post Market Clinical Follow-up (PMCF) is conducted to collect clinical and radiographic outcome information on patients suffering from intractable symptomatic cervical disc disease requiring 1- or 2-level reconstruction of the disc from C3-C7, after being treated with the Triadyme-C polycrystalline diamond compact cervical disc replacement.

ELIGIBILITY:
Inclusion Criteria:

1. 1- or 2-level cTDR surgery between C3 and C7
2. Age ≥ 18 years
3. Skeletally mature patient
4. Patient suffers from intractable symptomatic cervical disc disease (SCDD) with neck or arm (radicular) pain and/or a functional/neurological deficit
5. At least one of the following conditions must be present and confirmed by radiographic (CT, MRI, x-ray, etc.) studies: herniated nucleus pulposus, spondylosis (indicated by the presence of osteophytes), or loss of disc height.
6. At least six weeks of non-operative treatment for SCDD has been tried and failed prior to implantation
7. Psychosocially, mentally, and physically able to fully comply with the clinical protocol and willing to adhere to follow-up schedule and requirements.
8. Patient signed Informed Consent

Exclusion Criteria:

1. Active systemic infection or infection localized to the site of implantation
2. Allergy or sensitivity to the implant materials
3. Osteoporosis, defined as a Dual-energy X-ray Absorptiometry (DXA) bone mineral density T-score equal to or less than -2.5
4. Marked cervical instability on radiographs (e.g., radiographic signs of subluxation greater than 3.5 mm or angulation of the disc space more than 11 degrees greater than adjacent segments)
5. Severe spondylosis characterized by bridging osteophytes or an absence of motion (less than 2 degrees)
6. Significant cervical anatomical deformity or compromised vertebral bodies at the index level (e.g. ankylosing spondylitis, rheumatoid arthritis, or compromise due to current or past trauma)
7. Significant kyphotic deformity or significant reversal of lordosis
8. Previous cervical spinal surgery, other than discectomy at the levels to be operated on
9. Use of any spinal implant other than Triadyme-C
10. Adiposity, severe obesity (BMI > 40 kg/m2)
11. Patient who takes immunosuppressive or long-term steroid use
12. Fever
13. Systemic or metabolic illnesses (i.e. disease of bone-metabolism, insulin-dependent diabetes ...)
14. Patient who is suffering from rheumatoid or other inflammatory joint disease
15. Patient with any known active malignancy within the last 2 years
16. Any medical or surgical condition that could preclude the potential success of the implantation
17. Psychosocial issues; lack of co-operation by the patient, drug abuse or alcoholism
18. Unwillingness or inability of the patient to follow the instructions for postoperative treatment or with the follow-up evaluation schedule
19. Female patient who is pregnant or plans to become pregnant during the course of the study
20. Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic of selected spine centers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2020-05 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | 2 years postoperative
  Clinical outcome is measured by the Neck Disability Index (NDI) as published by Vernon et. al.. The primary endpoint of the study will be the mean total NDI at the 2 year postoperative assessment.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) on neck pain | 2 years postoperative
  The Visual Analogue Scale (VAS) represents the subject's intensity of neck pain during the last week measured on a line of 10 cm length, stretching from 'no pain (0 cm) to 'pain as bad as it could be' (10 cm).
Visual Analogue Scale (VAS) on arm pain | 2 years postoperative
  The VAS represents the subject's intensity of pain experienced in the pain-dominant arm during the last week measured on a line of 10 cm length, stretching from 'no pain (0 cm) to 'pain as bad as it could be' (10 cm).
Rate of device failure | 2 years postoperative
  Failure rate is based on the number of subjects whose radiographs, MRIs and/or CTs showed one or more device failures during the 2 year follow-up period after implantation divided by the total number of patients with 2 year radiographs or earlier failures.
Rate of subsequent surgical interventions | 2 years postoperative
  The following subsequent surgical intervention rates at index level are secondary study endpoints
  * removal
  * revision
  * reoperation
  * supplemental fixation
  Each subsequent surgical intervention rate is based on the number of subjects who showed one or more surgical interventions at index level per category during the 2 year follow-up period after implantation divided by the total number of patients with 2 year results or earlier subsequent surgical interventions.
Range of motion at index level | 2 years postoperative
  Range of motion (ROM) at index level means the degree of flexion/extension motion in the replaced segment. It is measured along the endplates according to the technique of Cobb in degrees in the sagittal plane on active lateral flexion and extension radiographs. ROM is defined as the difference of endplate alignment (Cobb angle) in maximum active flexion and maximum active extension per follow-up examination.
Rate of subsequent surgical interventions at symptomatic adjacent levels | 2 years postoperative
  The rate of subsequent surgical interventions at symptomatic adjacent levels is based on the number of subjects who underwent subsequent surgery to treat progressive adjacent segment disease during the 2 year follow-up period after implantation divided by the total number of patients with 2 year results or earlier adjacent subsequent surgical interventions.

OTHER OUTCOMES:
Adverse Events | 2 years postoperative
  Reporting of AE (adverse device effects (ADE) / procedure related AEs / other AEs) and by seriousness (serious AE (SAE) / non-serious AE) and intensity (mild / moderate / severe) is performed by the Principal Investigator based upon all reported adverse events.
Change in postoperative disc height at index level | 2 years postoperative
  Postoperative disc height at index level means the average disc height at the instrumented level. Therefore the anterior and posterior height will be measured from neutral lateral radiographs according to the radiographic protocol. Average height is calculated as the average of the corresponding anterior and posterior heights. Correction of magnification is performed for all distances measured according to the radiographic protocol.
Heterotopic ossification (HO) at index level | 2 years postoperative
  HO is evaluated according to McAfee et al.
Neurological status | 2 years postoperative
  The patient's neurological function is recorded preoperatively and at all postoperative follow-ups. The assessment includes motor, sensory and reflex evaluations by dermatome.
Patient's work status | 2 years postoperative
  The patient's work status is recorded by the patient preoperatively and at all postoperative follow-ups. It is documented by the following categories:
  * working
  * not working due to neck disability
  * not working for reasons other than neck disability
Patient's satisfaction | 2 years postoperative
  A VAS represents the patient's satisfaction with the outcome of the cTDR during the last week measured on a line of 10 cm length, stretching from 'extremely satisfied' (0 cm) to 'extremely dissatisfied' (10 cm).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Spiller, MD, Principal Investigator — Stenum Ortho GmbH
Locations (4):
- Germany (4):
  - Orth.med, Kümmersbruck, Bavaria
  - STENUM Ortho GmbH, Ganderkesee, Lower Saxony
  - Klinikum der Universität Rostock Abteilung für Neurochirurgie, Rostock, Mecklenburg-Vorpommern
  - Charité Universitätsmedizin Berlin Klinik für Unfall- und Wiederherstellungschirurgie, Berlin

IPD SHARING:
Plan to Share IPD: No